CLINICAL TRIAL: NCT06022068
Title: Evaluating Rapamycin Treatment in Alzheimer's Disease Using Positron Emission Tomography (ERAP)
Brief Title: Evaluating Rapamycin Treatment in Alzheimer's Disease Using Positron Emission Tomography
Acronym: ERAP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Jonas Svensson, MD, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-00611-01
Record Dates: First submitted 2023-08-15; First posted 2023-09-01 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rapamycin (Experimental): Sirolimus tablets will be administered orally, 7 mg once per week during 26 weeks
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — 7 mg taken once per week during 26 weeks.
  Other Names: Rapamycin

SUMMARY:
This single-center, uncontrolled pilot study aims to evaluate the efficacy, safety, and tolerability of six months of intermittently dosed oral rapamycin (sirolimus) in subjects with early-stage Alzheimer's disease.

Fifteen participants will be recruited. Following a set of baseline measurements, all participants will receive a weekly oral dose of 7 mg rapamycin for six months. Participants will be continuously monitored for safety and side effects. At the termination of the treatment, follow-up measurements will be taken.

The primary endpoint will be change in cerebral glucose metabolism, measured using 18F labeled fluorodeoxyglucose ([18F]FDG) positron emission tomography (PET).

In addition to the registered outcome measures this pilot trial will explore the feasibility of acquiring data on the effect of sirolimus treatment on age-related tissue changes in the body using a variety of imaging modalities, such as bone mineral density assessed using quantitative computed tomography, retinal structures assessed using optical coherence tomography, periodontal tissue assessed using MRI and FDG-PET, cardiac function assessed using MRI, vessel wall in large arteries using MRI and [18F]FDG PET.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of mild cognitive impairment (MCI), or dementia of Alzheimer's type
2. Amyloid positivity established with either amyloid positron emission tomography or cerebrospinal fluid analysis.
3. For subjects with dementia, the disease should be in an early stage, operationalized as:

   * Stage 4 (Mild dementia) or lower, according to the National Institute on Aging - Alzheimer's Association 2018 clinical staging criteria, AND
   * Clinical Dementia Rating Scale (CDR) global score of 1 or lower, AND
   * Montreal Cognitive Assessment (MoCA) score of ≥ 18 OR Rey Auditory Verbal Learning Test (RAVLT) >4 words after 30 minutes
4. Capable of giving, and has the capacity to give informed consent
5. Availability of a responsible study partner who can accompany the subject to all planned visits
6. Male or female between 50 and 80 years
7. Normal or clinically acceptable medical history, physical examination, and vital signs

Exclusion Criteria:

1. History of any major disease that may interfere with safe engagement in the intervention (especially severe liver or kidney disease, or uncontrolled diabetes).
2. Central nervous system infarct, infection, or focal lesions of clinical significance on MRI scans.
3. Fulfills any contraindication for the use of sirolimus as per the summary of product characteristics, including but not restricted to:

   * Current or planned medication with a strong inhibitor of CYP3A4 or P-gp
   * Current or planned medication with a strong inducer of CYP3A4 or P-gp
   * Other current medications with known serious interaction risks with sirolimus
   * Known allergy or hypersensitivity to sirolimus
4. Significant obesity
5. Untreated and clinically significant hyperlipidemia
6. Treatment with immunosuppressive medications within the last 90 days (topical and nasal corticosteroids and inhaled corticosteroids for asthma are permitted), or chemotherapeutic agents for malignancy within the last 3 years
7. Major surgery within 3 months prior to the planned start of sirolimus treatment, OR has major surgery planned during the period of the trial.
8. Use of experimental medications for Alzheimer's or any other investigational medication or device within 60 days. Participants who have been involved in a monoclonal antibody study are excluded unless it is known that they were receiving placebo in that trial

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
Change in cerebral glucose metabolism | From baseline to six months
  Cerebral glucose uptake measured through [18F]FDG positron emission tomography

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | From baseline to six months
  Safety and tolerability of intermittent sirolimus treatment
Change in Cerebrospinal fluid (CSF) concentration of amyloid beta 42 | From baseline to six months
  CSF biomarker for Alzheimers disease
Change in CSF concentration of phosphorylated tau | From baseline to six months
  CSF biomarker for Alzheimers disease
Change in CSF concentration of total tau | From baseline to six months
  CSF biomarker for Alzheimers disease
Change in cerebral blood flow | From baseline to six months
  Cerebral blood flow measured with MRI using arterial spin labeling
Area under the concentration versus time curve (AUC) of sirolimus | Tested at one occasion between baseline to six months
  Whole blood measurements of sirolimus concentration.
Peak Plasma Concentration (Cmax) of sirolimus | Tested at one occasion between baseline to six months
  Whole blood measurements of sirolimus concentration.
Trough Plasma Concentration (Cmin) of sirolimus | Tested at one occasion between baseline to six months
  Whole blood measurements of sirolimus concentration.
Change in Montreal Cognitive Assessment (MoCA) rating | From baseline to six months
  Cognition assessed using the MoCA rating scale (0-30 points, higher scores indicating better cognitive performance)

OTHER OUTCOMES:
Change in composite z-score of neuropsychological tests | From baseline to six months
  Cognition assessed with a composite score of the following tests: Rey Auditory Verbal Learning Test; Rey-Osterrieth Complex Figure; Hagman test; Trail Making Test A + B; Wechsler Adult Intelligence Scale (subtest to assess processing speed/attention). A composite score will be calculated using z-score approach..
Change in concentration of neurofilament light in CSF | From baseline to six months
  Neuronal damage assessed using concentraion of neurofilament light in CSF.
Change in quotient of albumin concentration in serum and CSF | From baseline to six months
  Blood-brain barrier integrity assessed using quotient of concentration albumin in serum and CSF
Change in hand-grip strength | From baseline to six months
  Measured using a hand-grip dynamometer
Change in chair stand test | From baseline to six months
  Number of completed chair stands in 30 seconds
Change in walking speed | From baseline to six months
  Timed 10-metre dual task walking test
Change in ratio of CSF concentration of amyloid beta 42 and 40 | From baseline to six months
  CSF biomarker for Alzheimers disease

CONTACTS AND LOCATIONS:
Overall Officials: Pontus Plavén Sigray, PhD, Study Director — Karolinska Institutet; Jonas Svensson, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital Memory clinic, Solna, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
We aim to share pseudonymized individual participant data that underlie results in a publication in accordance with institutional regulations.

REFERENCES:
- [Derived] Wallgren HA, Kivipelto M, Plaven-Sigray P, Svensson JE. Pharmacokinetic analysis of intermittent rapamycin administration in early-stage Alzheimer's Disease. Geroscience. 2025 Oct 5. doi: 10.1007/s11357-025-01911-3. Online ahead of print. PMID 41046300
- [Derived] Svensson JE, Bolin M, Thor D, Williams PA, Brautaset R, Carlsson M, Sorensson P, Marlevi D, Spin-Neto R, Probst M, Hagman G, Moren AF, Kivipelto M, Plaven-Sigray P. Evaluating the effect of rapamycin treatment in Alzheimer's disease and aging using in vivo imaging: the ERAP phase IIa clinical study protocol. BMC Neurol. 2024 Apr 4;24(1):111. doi: 10.1186/s12883-024-03596-1. PMID 38575854